CLINICAL TRIAL: NCT01041105
Title: Laparoscopic Revision Roux-en-Y Gastric Bypass Surgery After Previous Anti-rflux Surgery: Intermediate Results
Brief Title: Gastric Bypass After Previous Anti-reflux Surgery
Acronym: RYGBafterARS
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Kelvin D Higa, MD; FACS; FASMBS; Professor of Surgery, University of California San Francisco, UCSF Fresno / ALSA Medical Group, Inc. Minimally Invasive Surgery Program
Other Study IDs: CMC IRB No. 2008086; U1111-1112-9919 (Other: World Health Organization, Universal Trial Number)
Record Dates: First submitted 2009-12-26; First posted 2009-12-31 (Estimated); Last update posted 2010-01-01 (Estimated); Status verified 2009-12

CONDITIONS: Clinically Severe Obesity; Gastroesophageal Reflux Disease
Keywords: Obesity; Gastroesophageal Reflux Disease; Nissen funduplication; Antireflux surgery; Revisional Gastric Bypass; Re-operative bariatric surgery; Bariatric surgery; Nissen; Conversion of Nissen to Gastric Bypass
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Gastric bypass after previous Nissen

SUMMARY:
The goal of this study is to describe the clinical presentation, indications, and operative treatment as well as assess the morbidity, mortality, and overall performance of revisional Roux-en-Y gastric bypass (RYGB) after either failed or functional antireflux surgery "ARS" in obese patients. With such information, we hope to determine which features might assist us in advancing our knowledge about Gastro-Esophageal Reflux Disease "GERD", the best option for primary ARS, and mechanisms of failure in the obese population as well as in identifying predictors of outcome after revisional surgery in this population.

DETAILED DESCRIPTION:
The epidemic of overweight and obesity in the United States of America along with its comorbidities continues to expand. Bariatric surgery has demonstrated to be the most effective and sustained method to control severe obesity and its comorbidities. For instance, type 2 diabetes mellitus was completely resolved in 76.8 percent, systemic arterial hypertension was resolved in 61.7 percent, dyslipidemia improved in 70 percent, and obstructive sleep apnea-hypopnea syndrome was resolved in 85.7 percent. Furthermore, bariatric surgery significantly increases life expectancy (89 percent) and decreases overall mortality (30-40 percent), particularly deaths from diabetes, heart disease, and cancer. Lastly, preliminary evidence about downstream savings associated with bariatric surgery offset the initial costs in 2 to 4 years.

Since 1998, there has been a substantially progressive increase in bariatric surgery. In 2005, the American Society of Metabolic and Bariatric Surgery "ASMBS" reported that 81 percent of bariatric procedures were approached laparoscopically. 205,000 people, in 2007, had bariatric surgery in the United States from which approximately 80 percent of these were Gastric Bypass. Moreover, there is a mismatch between eligibility and receipt of bariatric surgery with just less than 1 percent of the eligible population being treated for morbid obesity through bariatric surgery. Along with the increasing number of elective primary weight loss procedures, up to 20 percent of post RYGB patients cannot sustain their weight loss beyond 2 to 3 years after the primary bariatric procedure. Thus, revisional surgery for poor weight loss and re-operations for technical or mechanical complications will rise in a parallel manner.

Three systematic reviews and meta-analysis have examined the association between obesity (BMI >30kg/m2) and several GERD-related disorders, including 1) GERD symptoms, 2) erosive esophagitis "EE", and 3) esophageal adenocarcinoma "EA". Obesity is associated with a 1.5-to-2-fold increased risk of GERD symptoms and EE and a 2- to 2.5-fold increased risk of EA. In two large case-control studies, abdominal diameter (waist-hip ratio), but not BMI, is an independent risk factor for another GERD-related disorder, Barrett´s esophagus "BE".

Current pathophysiological mechanisms of GERD in the obese encompass the following. 1) Mechanical: I) increased intra-gastric pressure: increased intra-peritoneal and abdominal wall fat mass increases the intra-abdominal and peri-gastric pressures with subsequent increased gastroesophageal pressure gradient "GEPE" with augmented esophageal acid exposure. Each BMI unit increase corresponds to a 10 percent increase in intra-gastric pressure. II) Hiatal Hernia: "HH" disrupts the integrity of the sphincter mechanisms and prolongs esophageal acid clearance. Thin, normal, overweight, and obese subjects have a 1.0, 1.9, 2.5, and 4.2 risk of having HH compared to thin subjects, respectively. 2) Motility: I) Increased Transient LES Relaxation "TLESR" are associated with acid reflux during the postprandial period, especially during inspiration. II) Low LES basal pressure: Increased prevalence of abnormally low LES basal pressure in the overweight and obese in comparison to the normoweight subject. III) Esophageal motility abnormality: Jaffin et al, with esophageal manometry, reported 61 percent of patients with altered esophageal motility from which 59 percent had altered visceral pain perception (asymptomatic). IV) Delayed gastric emptying: mostly associated with one of its major comorbidities, diabetes mellitus. 3) Esophageal sensitivity: Mercer et al., with a Bernstein test, found a significant difference between normoweight and obese subjects without clinical evidence of GERD (0 percent vs. 86 percent, respectively) for esophageal hypersensitivity. 4) Hormonal: mostly mediated by estrogen and adiponectin. 5) Environmental (Diet): high-fat, saturated fatty acids, high-cholesterol, and high caloric density diets have been associated with the highest likelihood of perceiving an acid reflux event; fat may confer its sensory effect by activating pain facilitatory pathways or by deactivating pain inhibitory pathways.

The most recent data is not conclusive on whether increased BMI affects acid-suppressive therapy for GERD. However, MacDougall et al. found that increased BMI was significantly associated with long-term acid suppression therapy. This can be explained based on either a higher prevalence of factors that predispose overweight and obese subjects to severe GERD, such as HH, greater GEPG, increased number of TLESR, or standard doses of PPI´s are suboptimal for patients with increased BMI and GERD.

Broad indications for antireflux surgery include: 1) Reflux of food associated with HH, 2) despite successful medical treatment or after poor or moderate symptom control on optimized PPI therapy, patient opts for surgery, and 3) Complicated GERD without including severe dysplasia.

Available traditional ARS are either 1) fundoplication, which is the most commonly performed procedure and can be partial -Toupet, Dor- or complete -Nissen-, or other procedures with limited use such as 2) Hill operation, 3) pyloroplasty, 4) vagotomy with antrectomy, and 5) duodenal switch.

Long-term control of typical symptoms after primary laparoscopic Nissen fundoplication "LNF", in properly selected patients and with an experienced surgical team, is attained in more than 90 percent of patients confirming that LNF is the gold standard for the treatment of severe GERD.

In a cohort study of 166 patients followed for 11 years, Smith et al found preoperative response to acid-reducing medication, typical symptoms, and BMI < 35 Kg/m2 to predict successful outcome. However, HH size, normal 24-hour pH score, age > 50 years, female gender, and prior abdominal surgery that previous studies found to be associated with poor outcomes were not corroborated by this study. Other risk factors for failure are short esophagus, HH greater than 3 cm, and diaphragmatic stressors such as retching, sports of weight lifting, and high-speed motor vehicle accident among others.

Another study found increased BMI to be a predictor of poor outcome. Perez et al, in a retrospective cohort analysis of 224 patients undergoing LNF and transthoracic ARS, found a significantly increased recurrence rate of GERD in obese and overweight compared to normoweight patients, regardless of procedure type.

In contrast, a cohort study of 257 consecutive patients undergoing LNF, D´Alessio et al analyzed outcomes based on BMI (< 25, 25-30, and >30 kg/m2); No significant differences in symptom scores and clinical success rates were found among the different subsets. However, mean BMI for obese patients was 33 kg/m2 (obesity class I) and only three patients were >35 kg/m2.

Regardless of contradictory data about LNF efficacy in obesity, several studies have shown the effectiveness of RYGB for GERD in morbidly obese patients by symptoms, endoscopic findings, manometry and pH-metry results, and endoscopic biopsy-histopathology.

There are four retrospective cohort studies assessing mostly early outcomes after converting ARS to RYGB. First, Sarr et al analyzed 19 patients that underwent open conversion to RYGB. Next, Ikramuddin et al described the anatomic findings for fundoplication failure after the laparoscopic conversion to RYGB of 11 patients. Lastly, with seven patients each, Raftopoulos et al and Donnelly et al reported feasibility with a high morbidity rate as well.

In summary, there is little information about what is the best primary ARS and the best revisional strategy to address intractable or severe reflux after failed fundoplication in the obese population. Also, there is lack of data about the best revisional procedure to address obesity in the patient status post functional or competent ARS. With this pilot retrospective study, we will advance our knowledge and along with the existing literature, we will draw preliminary clinical recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Status post, either open or laparoscopic, primary Nissen fundoplication with all the following requirements:

  * Met NIH criteria for bariatric surgery
  * With functional or failed antireflux surgery (Nissen fundoplication)
  * Laparoscopic approach for revisional surgery

Exclusion Criteria:

* Any other type of revisional bariatric procedure
* Nonstandard revisional RYGB surgery
* Open approach for revision surgery
* Missing records and/or unreachable patients with scant information for analysis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who underwent laparoscopic Roux-en-Y gastric bypass (RYGB) after a previous functional or failed anti-reflux procedure and met National Institutes of Health criteria for bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Morbidity and mortality | at discharge, 1 week, 3 weeks, 8 weeks, 3 months, 6 months, 1 year and annually thereafter for up to 4 years
Remission or improvement of GERD-related symptoms | 6 months, 1 year and annually thereafter for up to 4 years
Weight loss expressed as Body Mass Index and Percentage of excess weight loss | 6 months, 1 year, and annually thereafter for up to 4 years

SECONDARY OUTCOMES:
Remission or improvement of comorbidities | 6 months, 1 year, and annually thereafter for up to 4 years
Length of operative time which is defined as the time duration of operation measured in minutes from the first skin incision to the final closure of the skin incision | It is measured in minutes from the first skin incision to the final closure of the skin incision at the time of revisional surgery under study. It is a transoperative measure of outcome of the surgery under study
Length of Hospital Stay which is a measured of surgical recovery quantified and reported in days. It is a hospital pre-discharge traditional measure of outcome. | It is measured in days from the admission date to the discharge date for the hospitalization pertaining to revisional surgery under study

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Tercero, MD, Study Director — Research Associate, University of California San Francisco; Kelvin D Higa, MD, Principal Investigator — Professor of Surgery, University of California San Francisco
Locations (1):
- UCSF Fresno Center for Medical Education and Research, Fresno, California, United States

REFERENCES:
- [Background] Higa KD, Boone KB, Ho T, Davies OG. Laparoscopic Roux-en-Y gastric bypass for morbid obesity: technique and preliminary results of our first 400 patients. Arch Surg. 2000 Sep;135(9):1029-33; discussion 1033-4. doi: 10.1001/archsurg.135.9.1029. PMID 10982506
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- [Background] McTigue KM, Harris R, Hemphill B, Lux L, Sutton S, Bunton AJ, Lohr KN. Screening and interventions for obesity in adults: summary of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2003 Dec 2;139(11):933-49. doi: 10.7326/0003-4819-139-11-200312020-00013. PMID 14644897
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Christou NV, Sampalis JS, Liberman M, Look D, Auger S, McLean AP, MacLean LD. Surgery decreases long-term mortality, morbidity, and health care use in morbidly obese patients. Ann Surg. 2004 Sep;240(3):416-23; discussion 423-4. doi: 10.1097/01.sla.0000137343.63376.19. PMID 15319713
- [Background] Adams TD, Gress RE, Smith SC, Halverson RC, Simper SC, Rosamond WD, Lamonte MJ, Stroup AM, Hunt SC. Long-term mortality after gastric bypass surgery. N Engl J Med. 2007 Aug 23;357(8):753-61. doi: 10.1056/NEJMoa066603. PMID 17715409
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Cremieux PY, Buchwald H, Shikora SA, Ghosh A, Yang HE, Buessing M. A study on the economic impact of bariatric surgery. Am J Manag Care. 2008 Sep;14(9):589-96. PMID 18778174
- [Background] Santry HP, Gillen DL, Lauderdale DS. Trends in bariatric surgical procedures. JAMA. 2005 Oct 19;294(15):1909-17. doi: 10.1001/jama.294.15.1909. PMID 16234497
- [Background] Flum DR, Khan TV, Dellinger EP. Toward the rational and equitable use of bariatric surgery. JAMA. 2007 Sep 26;298(12):1442-4. doi: 10.1001/jama.298.12.1442. No abstract available. PMID 17895461
- [Background] Meguid MM, Glade MJ, Middleton FA. Weight regain after Roux-en-Y: a significant 20% complication related to PYY. Nutrition. 2008 Sep;24(9):832-42. doi: 10.1016/j.nut.2008.06.027. PMID 18725080
- [Background] Nguyen NT. Reoperations and revisions in bariatric surgery. Surg Endosc. 2007 Nov;21(11):1907-8. doi: 10.1007/s00464-007-9572-6. Epub 2007 Sep 8. No abstract available. PMID 17828427
- [Background] Hampel H, Abraham NS, El-Serag HB. Meta-analysis: obesity and the risk for gastroesophageal reflux disease and its complications. Ann Intern Med. 2005 Aug 2;143(3):199-211. doi: 10.7326/0003-4819-143-3-200508020-00006. PMID 16061918
- [Background] Corley DA, Kubo A. Body mass index and gastroesophageal reflux disease: a systematic review and meta-analysis. Am J Gastroenterol. 2006 Nov;101(11):2619-28. doi: 10.1111/j.1572-0241.2006.00849.x. Epub 2006 Sep 4. PMID 16952280
- [Background] Kubo A, Corley DA. Body mass index and adenocarcinomas of the esophagus or gastric cardia: a systematic review and meta-analysis. Cancer Epidemiol Biomarkers Prev. 2006 May;15(5):872-8. doi: 10.1158/1055-9965.EPI-05-0860. PMID 16702363
- [Background] Corley DA, Kubo A, Levin TR, Block G, Habel L, Zhao W, Leighton P, Quesenberry C, Rumore GJ, Buffler PA. Abdominal obesity and body mass index as risk factors for Barrett's esophagus. Gastroenterology. 2007 Jul;133(1):34-41; quiz 311. doi: 10.1053/j.gastro.2007.04.046. Epub 2007 Apr 25. PMID 17631128
- [Background] Edelstein ZR, Farrow DC, Bronner MP, Rosen SN, Vaughan TL. Central adiposity and risk of Barrett's esophagus. Gastroenterology. 2007 Aug;133(2):403-11. doi: 10.1053/j.gastro.2007.05.026. Epub 2007 May 21. PMID 17681161
- [Background] Fass R. The pathophysiological mechanisms of GERD in the obese patient. Dig Dis Sci. 2008 Sep;53(9):2300-6. doi: 10.1007/s10620-008-0411-y. Epub 2008 Jul 29. PMID 18663576
- [Background] Jacobson BC. Body mass index and the efficacy of acid-mediating agents for GERD. Dig Dis Sci. 2008 Sep;53(9):2313-7. doi: 10.1007/s10620-008-0414-8. Epub 2008 Jul 16. PMID 18629639
- [Background] Morgenthal CB, Shane MD, Stival A, Gletsu N, Milam G, Swafford V, Hunter JG, Smith CD. The durability of laparoscopic Nissen fundoplication: 11-year outcomes. J Gastrointest Surg. 2007 Jun;11(6):693-700. doi: 10.1007/s11605-007-0161-8. PMID 17562117
- [Background] Bammer T, Hinder RA, Klaus A, Klingler PJ. Five- to eight-year outcome of the first laparoscopic Nissen fundoplications. J Gastrointest Surg. 2001 Jan-Feb;5(1):42-8. doi: 10.1016/s1091-255x(01)80012-3. PMID 11309647
- [Background] Dallemagne B, Weerts J, Markiewicz S, Dewandre JM, Wahlen C, Monami B, Jehaes C. Clinical results of laparoscopic fundoplication at ten years after surgery. Surg Endosc. 2006 Jan;20(1):159-65. doi: 10.1007/s00464-005-0174-x. Epub 2005 Dec 7. PMID 16333553
- [Background] Morgenthal CB, Lin E, Shane MD, Hunter JG, Smith CD. Who will fail laparoscopic Nissen fundoplication? Preoperative prediction of long-term outcomes. Surg Endosc. 2007 Nov;21(11):1978-84. doi: 10.1007/s00464-007-9490-7. Epub 2007 Jul 11. PMID 17623236
- [Background] O'Boyle CJ, Watson DI, DeBeaux AC, Jamieson GG. Preoperative prediction of long-term outcome following laparoscopic fundoplication. ANZ J Surg. 2002 Jul;72(7):471-5. doi: 10.1046/j.1445-2197.2002.02455.x. PMID 12123502
- [Background] Power C, Maguire D, McAnena O. Factors contributing to failure of laparoscopic Nissen fundoplication and the predictive value of preoperative assessment. Am J Surg. 2004 Apr;187(4):457-63. doi: 10.1016/j.amjsurg.2003.12.034. PMID 15041491
- [Background] Campos GM, Peters JH, DeMeester TR, Oberg S, Crookes PF, Tan S, DeMeester SR, Hagen JA, Bremner CG. Multivariate analysis of factors predicting outcome after laparoscopic Nissen fundoplication. J Gastrointest Surg. 1999 May-Jun;3(3):292-300. doi: 10.1016/s1091-255x(99)80071-7. PMID 10481122
- [Background] Perez AR, Moncure AC, Rattner DW. Obesity adversely affects the outcome of antireflux operations. Surg Endosc. 2001 Sep;15(9):986-9. doi: 10.1007/s004640000392. Epub 2001 Jun 12. PMID 11443428
- [Background] D'Alessio MJ, Arnaoutakis D, Giarelli N, Villadolid DV, Rosemurgy AS. Obesity is not a contraindication to laparoscopic Nissen fundoplication. J Gastrointest Surg. 2005 Sep-Oct;9(7):949-54. doi: 10.1016/j.gassur.2005.04.019. PMID 16137590
- [Background] Frezza EE, Ikramuddin S, Gourash W, Rakitt T, Kingston A, Luketich J, Schauer P. Symptomatic improvement in gastroesophageal reflux disease (GERD) following laparoscopic Roux-en-Y gastric bypass. Surg Endosc. 2002 Jul;16(7):1027-31. doi: 10.1007/s00464-001-8313-5. Epub 2002 May 3. PMID 11984683
- [Background] Smith SC, Edwards CB, Goodman GN. Symptomatic and clinical improvement in morbidly obese patients with gastroesophageal reflux disease following Roux-en-Y gastric bypass. Obes Surg. 1997 Dec;7(6):479-84. doi: 10.1381/096089297765555205. PMID 9730504
- [Background] Patterson EJ, Davis DG, Khajanchee Y, Swanstrom LL. Comparison of objective outcomes following laparoscopic Nissen fundoplication versus laparoscopic gastric bypass in the morbidly obese with heartburn. Surg Endosc. 2003 Oct;17(10):1561-5. doi: 10.1007/s00464-002-8955-y. Epub 2003 Jul 21. PMID 12874685
- [Background] Houghton SG, Romero Y, Sarr MG. Effect of Roux-en-Y gastric bypass in obese patients with Barrett's esophagus: attempts to eliminate duodenogastric reflux. Surg Obes Relat Dis. 2008 Jan-Feb;4(1):1-4; discussion 4-5. doi: 10.1016/j.soard.2007.10.003. Epub 2007 Dec 19. PMID 18069070
- [Background] Houghton SG, Nelson LG, Swain JM, Nesset EM, Kendrick ML, Thompson GB, Murr MM, Nichols FC, Sarr MG. Is Roux-en-Y gastric bypass safe after previous antireflux surgery? Technical feasibility and postoperative symptom assessment. Surg Obes Relat Dis. 2005 Sep-Oct;1(5):475-80. doi: 10.1016/j.soard.2005.07.004. Epub 2005 Aug 31. PMID 16925273
- [Background] Kellogg TA, Andrade R, Maddaus M, Slusarek B, Buchwald H, Ikramuddin S. Anatomic findings and outcomes after antireflux procedures in morbidly obese patients undergoing laparoscopic conversion to Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2007 Jan-Feb;3(1):52-7; discussion 58-9. doi: 10.1016/j.soard.2006.08.011. Epub 2006 Nov 20. PMID 17116426
- [Background] Raftopoulos I, Awais O, Courcoulas AP, Luketich JD. Laparoscopic gastric bypass after antireflux surgery for the treatment of gastroesophageal reflux in morbidly obese patients: initial experience. Obes Surg. 2004 Nov-Dec;14(10):1373-80. doi: 10.1381/0960892042583950. PMID 15603654
- [Background] Zainabadi K, Courcoulas AP, Awais O, Raftopoulos I. Laparoscopic revision of Nissen fundoplication to Roux-en-Y gastric bypass in morbidly obese patients. Surg Endosc. 2008 Dec;22(12):2737-40. doi: 10.1007/s00464-008-9848-5. Epub 2008 Mar 25. PMID 18363066
- [Background] Donnelly PE, Salgado JJ, Gagne DD, et al. Efficacy of laparoscopic Roux-en-Y gastric bypass (LRYGB) in obese patients with a previous fundoplication. Surg Obes Relat Dis 2007;3: 299-344.
- [Background] Ikramuddin S. Surgical management of gastroesophageal reflux disease in obesity. Dig Dis Sci. 2008 Sep;53(9):2318-29. doi: 10.1007/s10620-008-0415-7. Epub 2008 Jul 29. PMID 18663575
- See also: "Click here for more information about the department sponsor´s web site" — http://www.fresno.ucsf.edu/surgery/